CLINICAL TRIAL: NCT00157326
Title: A Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study Evaluating the Efficacy and Safety of Tadalafil (5mg and 20mg) Administered Once Daily to Subjects With Mild to Moderate Hypertension
Brief Title: Tadalafil in Subjects With Mild to Moderate Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10077; H6D-MC-LVGU
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2007-10

CONDITIONS: Hypertension
Keywords: High Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — Tadalafil

INTERVENTIONS:
Drug: tadalafil
  Other Names: LY450190; Cialis; IC351

SUMMARY:
Purpose: The primary objective of this study is to evaluate the efficacy and safety of tadalafil when administered once daily at doses of 5 and 20 mg to adult subjects for 8 weeks with mild to moderate hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented medical history of hypertension.
* Have cuff seated diastolic blood pressure values greater than or equal to 95 and less than or equal to 104 mm at study entry
* Have a negative serum pregnancy test at the time of enrollment and agree to use two medically reliable methods of contraception until study completion, if female is of child-bearing potential, between menarche and 1 year post menopause and not surgically sterilized.
* Are able to comply with study procedures and visits

Exclusion Criteria:

* Have resistant hypertension or systolic hypertension.
* Are obese, defined as having body mass index (BMI) greater than or equal to 35.
* Are females who are pregnant or breast feeding.
* Have a history of severe renal insufficiency or significant thyroid, renal or hepatic disease.
* Have a glycosylated hemoglobin A1c (HbA1c) greater than or equal to 10% during the screening period.
* Have significant anemia.
* Have a significant or unstable cardiac history such as history of heart attack, unstable angina, or stroke within 6 months of study entry, history of angina that was treated with long- or short-acting nitrates within 90 days of study entry, history of coronary artery bypass graft surgery or cardiac angioplasty within 90 days of study entry, history of abnormal heart rhythms such as sick sinus syndrome or 2nd- or 3rd-degree AV block, chronic atrial fibrillation or recurrent atrial tachyarrhythmia, a history of recurrent ventricular tachycardia, or symptomatic bradycardia, a history of sudden cardiac arrest.
* Have symptomatic heart failure requiring treatment, or significant disease of the heart valves.
* Have been treated for severe asthma, bronchospasm, or COPD within 3 months of study entry.
* Have severe peripheral vascular disease.
* Have a documented diagnosis of sleep apnea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2005-09; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
The primary efficacy measurement of this study is the mean change after 8 weeks of treatment from baseline in cuff seated trough diastolic blood pressure, cuff seated systolic blood pressures and automated blood pressure monitoring

SECONDARY OUTCOMES:
Safety will be assessed by evaluating all reported adverse events and changes in clinical laboratory values, ECGs, and vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bothell, Washington, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com